CLINICAL TRIAL: NCT01752036
Title: Phase II Study of Post-Operative Stereotactic Radiosurgery for Solid Tumor Spine Metastases
Brief Title: Radiotherapy for Solid Tumor Spine Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J12133; NA_00080433 (Other: JHMIRB)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumor Spine Metastases
Keywords: stereotactic radiotherapy; SRS
MeSH Terms: interventions — Postoperative Period; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Post-Operative Stereotactic Radiosurgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Other): Post-Operative Stereotactic Radiosurgery
  Interventions: Radiation: Post-operative, Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Post-operative, Stereotactic Body Radiation Therapy (SBRT) — All participants received SBRT at 600 cGy x 5 fractions

SUMMARY:
Although it is being increasingly used off protocol, there is minimal data regarding the efficacy of stereotactic radiosurgery to the tumor bed following surgical resection of metastatic lesions to the spine. The primary objective of this study is to evaluate radiographic local recurrence in the tumor bed following stereotactic radiosurgery compared to the expected rate following conventional radiation therapy.

DETAILED DESCRIPTION:
This is a phase II trial evaluating the rate radiographic local recurrence following post-operative stereotactic radiosurgery boost in patients with metastatic solid malignancies with spine metastases status post resection. Patients will be treated with 600 cGy x 5 fractions to the tumor bed and then followed both clinically and radiographically to determine if local recurrence following this treatment is better than might be expected for conventional radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years
* Histologically proven solid tumor malignancy with metastasis to the spine. Diagnosis may be acquired from needle biopsy, cytology, or surgical biopsy or resection.
* Radiographic evidence of spinal metastasis is required and may be obtained from plain radiographs, radionuclide bone scans, computed tomography imaging, and magnetic resonance imaging. Other studies may be used with principal investigator approval.
* The patient must have undergone surgical resection resection (gross total, subtotal, or biopsy) of the spinal lesion(s) no more than 12 weeks prior to SRS treatment.
* Treating physician must deem that SRS is appropriate treatment for the metastatic spinal lesion(s).
* Each SRS target must be the equivalent of ≤3 vertebral levels
* The patient must have a Karnofsky Performance Score of 40 or greater
* If a woman is of child-bearing potential, a negative urine or serum pregnancy test must be demonstrated prior to treatment. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for up to 12 weeks following the study. Should a woman become pregnant or suspect she is pregnant while participating in this study she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation or radiosurgery to the involved level of the spine
* Spine disease from leukemia, lymphoma or myeloma
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, or other cancer from which the patient has been disease free for at least 1 year.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements will be excluded.
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use and acceptable method of birth control to avoid pregnancy for the entire study period and up to 12 weeks after the study are excluded. Male subjects must also agree to use effective contraception for the same period as above.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Redmond KJ, Sciubba D, Khan M, Gui C, Lo SL, Gokaslan ZL, Leaf B, Kleinberg L, Grimm J, Ye X, Lim M. A Phase 2 Study of Post-Operative Stereotactic Body Radiation Therapy (SBRT) for Solid Tumor Spine Metastases. Int J Radiat Oncol Biol Phys. 2020 Feb 1;106(2):261-268. doi: 10.1016/j.ijrobp.2019.10.011. Epub 2019 Oct 16. PMID 31628959

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 of the 35 enrolled participants received treatment.
Period: Overall Study
Arm/Group | Treatment
Started | 33
Completed | 31
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: 35 participants were enrolled and baseline data was collected on all 35. However, only 33 participants actually started treatment.
Arm/Group | Treatment
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 63 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiographic Recurrence at 12 Months
Description: To estimate the rate of radiographic local recurrence at 12 months in patients treated with a post-operative stereotactic radiosurgery boost for resected spine metastases.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Participants | 3

2. Primary Outcome: Time to Local Recurrence
Description: To estimate the time (in months) to radiographic local recurrence in patients treated with a post-operative stereotactic radiosurgery boost for resected spine metastases.
Time Frame: 1 year
Measure: Median (Full Range); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 31
months | 3.5 [3.4 to 5.8]

3. Secondary Outcome: Number of Participants Receiving Re-treatment
Description: To estimate the rate of re-treatment at 12 months in patients treated with a post-operative stereotactic radiosurgery boost for resected spine metastases
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Participants | 2

4. Secondary Outcome: Number of Participants With Symptomatic Recurrence
Description: To estimate the rate of symptomatic local recurrence at 12 months in patients treated with a post-operative stereotactic radiosurgery boost for resected spine metastases
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Participants | 31

5. Secondary Outcome: Number of Participants Experiencing Radiation Myelopathy
Description: Number of participants experiencing radiation myelopathy in patients treated with a post-operative stereotactic radiosurgery boost for resected spine metastases
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Participants | 0

6. Secondary Outcome: Number of Participants Experiencing Wound Dehiscence
Description: Number of participants treated with a post-operative stereotactic radiosurgery boost for resected spine metastases, experiencing wound dehiscence.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Participants | 0

7. Secondary Outcome: Time to Return to Chemotherapy
Description: Time in months to return to chemotherapy in patients treated with a post-operative stereotactic radiosurgery boost for resected spine metastases.
Time Frame: 1 year
Measure: Median (Full Range); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 31
months | 0.5 [0 to 9.4]

8. Secondary Outcome: Number of Participants With Radio-sensitive Tumors Who Had Symptomatic Local Recurrence
Description: To evaluate the post-treatment symptomatic local recurrence in patients with radio-sensitive tumors.
Time Frame: 1 year
Population: Only 3 participants had radio-sensitive tumors.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Events were defined by Radiation Therapy Oncology Group (RTOG) and European Organisation for Research and Treatment of Cancer (EORTC) criteria.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 2/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 31/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment (N=33)
Agitation (Psychiatric disorders) | 16/31
Akathisia (Psychiatric disorders) | 3/31
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3/31
Anemia (Blood and lymphatic system disorders) | 24/31
Anorexia (Psychiatric disorders) | 17/31
Anxiety (Psychiatric disorders) | 16/31
AST increased (Gastrointestinal disorders) | 4/31
Bloating (Gastrointestinal disorders) | 10/31
Chills rigors (General disorders) | 3/31
Concentration impairment (General disorders) | 9/31
Constipation (Gastrointestinal disorders) | 21/31
Cough (General disorders) | 8/31
Depression (Psychiatric disorders) | 18/31
Diarrhea (Gastrointestinal disorders) | 6/31
Dizziness (General disorders) | 8/31
Dry mouth (General disorders) | 12/31
Dyspepsia (Gastrointestinal disorders) | 10/31
Dyphagia (Nervous system disorders) | 4/31
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7/31
Edema extremities (Metabolism and nutrition disorders) | 3/31
Fatigue (General disorders) | 29/31
Gastritis (Gastrointestinal disorders) | 6/31
Headache (General disorders) | 6/31
Insomnia (General disorders) | 5/31
Localized edema (Metabolism and nutrition disorders) | 4/31
Lymphocyte count decreased (Blood and lymphatic system disorders) | 6/31
Lymphocytes absolute decreased (Blood and lymphatic system disorders) | 8/31
Malaise (General disorders) | 7/31
Nausea (Gastrointestinal disorders) | 17/31
Neuralgia (Musculoskeletal and connective tissue disorders) | 16/31
Pain (General disorders) | 6/31
Pain due to RT (Surgical and medical procedures) | 3/31
Platelet count decreased (Blood and lymphatic system disorders) | 6/31
Stomach pain (Gastrointestinal disorders) | 11/31
Tremor (Nervous system disorders) | 10/31
Weight loss (Metabolism and nutrition disorders) | 15/31
White blood cell count decreased (Blood and lymphatic system disorders) | 9/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT01752036/Prot_SAP_000.pdf